CLINICAL TRIAL: NCT06006949
Title: Roxadustat Combined With Luspatercept Versus Luspatercept Monotherapy in the Treatment of Refractory Myelodysplastic Syndrome With Ring Sideroblasts (MDS-RS): A Prospective Randomized Controlled Study
Brief Title: Roxadustat Combined With Luspatercept Versus Luspatercept Monotherapy in the Treatment of Refractory MDS-RS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bing Han, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Lus-2
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — roxadustat; luspatercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- roxadustat and luspatercept (Experimental): Luspatercept (1.0 mg/kg, subcutaneously injection every 3 weeks, adjusted according to blood pattern, up to 1.75mg/kg.
  Roxadustat (150mgqod) was administered for at least 6 months to evaluate efficacy.
  Hemoglobin ≥120g/L can be discontinued, and hemoglobin <120g/L can continue to use. Those who are effective will continue to be given the combination therapy until ineffective or intolerant.
  Interventions: Drug: Roxadustat; Drug: Luspatercept
- luspatercept (Experimental): Luspatercept (1.0 mg/kg, subcutaneously injection every 3 weeks, adjusted according to blood pattern, up to 1.75mg/kg.
  Luspatercept was given for at least 6 months to evaluate the efficacy. Hemoglobin ≥120g/L can be discontinued, and hemoglobin <120g/L can continue to use. Those who are effective will continue to be given the therapy until it is ineffective or intolerant
  Interventions: Drug: Luspatercept

INTERVENTIONS:
Drug: Roxadustat — Roxadustat (150 mgqod)
  Arms: roxadustat and luspatercept
Drug: Luspatercept — Luspatercept (1.0 mg/kg, subcutaneously injection every 3 weeks, adjusted according to blood pattern, up to 1.75mg/kg)

SUMMARY:
In a randomized controlled phase II/III clinical trial, 58% of patients with lower-risk MDS had at least a 50% reduction in red blood cell (RBC) transfusion units every 8 weeks after roxadustat treatment. In a randomized controlled phase III clinical trial, luspatercept significantly improved transfusion dependence in erythropoietin-stimulating agents (ESA)-refractory MDS-RS and improved hemoglobin response and quality of life, compared to placebo. This study aimed to evaluate the efficacy and safety of roxadustat combined with luspatercept versus luspatercept monotherapy in the treatment of refractory MDS-RS.

DETAILED DESCRIPTION:
Myelodysplastic neoplasms (MDS) are heterogeneous clonal disorders of stem cells that result in peripheral blood cytopenia and ineffective hematopoiesis, with the potential risk of the development of acute myeloid leukemia (AML). Most patients with myelodysplastic syndromes with ring sideroblasts (MDS-RS) are stratified into lower-risk groups by the revised International Prognostic Scoring System (IPSS). At present, the main therapies for MDS-RS are red blood cell and platelet transfusion, erythropoietin (EPO), androgen, and iron chelation therapy. Roxadustat can up-regulate transferrin receptors to increase iron absorption, up-regulate transferrin to promote iron transport, and down-regulate ferritin levels to indirectly improve iron absorption and transport, promote plasma iron entry into the bone marrow to generate red blood cells and promote the production of EPO in the physiological range. Luspatercept generally promotes advanced erythrocyte maturation by inhibiting the TGF-β/smad2/3 signaling pathway. In a randomized controlled phase II/III clinical trial, 58% of patients with lower-risk MDS had at least a 50% reduction in red blood cell (RBC) transfusion units every 8 weeks after roxadustat treatment. In a randomized controlled phase III clinical trial, luspatercept significantly improved transfusion dependence in erythropoietin-stimulating agents (ESA)-refractory MDS-RS and improved hemoglobin response and quality of life, compared to placebo. The aim of this study was to evaluate the efficacy and safety of roxadustat combined with luspatercept versus luspatercept monotherapy in the treatment of refractory MDS-RS. If it is proved that the combination of the two drugs is better than luspatercept monotherapy, it can quickly improve the anemia of refractory MDS-RS and improve the quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years old.
2. Patients with a definite diagnosis of MDS-RS and stratified as lower-risk according to IPSS-R.
3. After at least 6 weeks of rhEPO treatment, with hemoglobin<100g/L
4. Adequate hepatic functions with alanine transaminase (ALT)/aspartate. transaminase (AST) levels within 2 times of the normal upper limit and total bilirubin levels within 2 times of the normal upper limit.
5. ECOG≤2 with an expected life span of more than 6 months
6. Documented patient consent.

Exclusion Criteria:

1. Age <18 years old.
2. Complicated with active or uncontrolled infections.
3. Complicated with other malignancies.
4. Creatinine/transaminase ≥ 2 normal upper limit.
5. Complicated with myelofibrosis.
6. Pregnant or lactating women, or men with recent fertility needs
7. Allergic to luspatercept or excipients
8. Patients with history of polysorbate 80 allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
overall response rate (ORR) | 6 month
  Proportion of patients who achieved complete response, partial response and hematological response.

SECONDARY OUTCOMES:
transfusion indenpendence (TI) | 6 month
  Proportion of patients with transfusion dependence over 8 weeks
adverse event rate | 6 month
  Proportion of patients with adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arber DA, Orazi A, Hasserjian R, Thiele J, Borowitz MJ, Le Beau MM, Bloomfield CD, Cazzola M, Vardiman JW. The 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia. Blood. 2016 May 19;127(20):2391-405. doi: 10.1182/blood-2016-03-643544. Epub 2016 Apr 11. PMID 27069254
- [Background] Zheng Q, Yang H, Fu X, Huang Y, Wei R, Wang Y, Liu YN, Liu WJ. The efficacy and safety of roxadustat for anemia in patients with chronic kidney disease: a meta-analysis. Nephrol Dial Transplant. 2021 Aug 27;36(9):1603-1615. doi: 10.1093/ndt/gfaa110. PMID 33051677
- [Background] Gupta N, Wish JB. Hypoxia-Inducible Factor Prolyl Hydroxylase Inhibitors: A Potential New Treatment for Anemia in Patients With CKD. Am J Kidney Dis. 2017 Jun;69(6):815-826. doi: 10.1053/j.ajkd.2016.12.011. Epub 2017 Feb 24. PMID 28242135
- [Background] Crugliano G, Serra R, Ielapi N, Battaglia Y, Coppolino G, Bolignano D, Bracale UM, Pisani A, Faga T, Michael A, Provenzano M, Andreucci M. Hypoxia-Inducible Factor Stabilizers in End Stage Kidney Disease: "Can the Promise Be Kept?". Int J Mol Sci. 2021 Nov 22;22(22):12590. doi: 10.3390/ijms222212590. PMID 34830468
- [Background] Chen N, Hao C, Liu BC, Lin H, Wang C, Xing C, Liang X, Jiang G, Liu Z, Li X, Zuo L, Luo L, Wang J, Zhao MH, Liu Z, Cai GY, Hao L, Leong R, Wang C, Liu C, Neff T, Szczech L, Yu KP. Roxadustat Treatment for Anemia in Patients Undergoing Long-Term Dialysis. N Engl J Med. 2019 Sep 12;381(11):1011-1022. doi: 10.1056/NEJMoa1901713. Epub 2019 Jul 24. PMID 31340116
- [Background] Henry DH, Glaspy J, Harrup R, Mittelman M, Zhou A, Carraway HE, Bradley C, Saha G, Modelska K, Bartels P, Leong R, Yu KP. Roxadustat for the treatment of anemia in patients with lower-risk myelodysplastic syndrome: Open-label, dose-selection, lead-in stage of a phase 3 study. Am J Hematol. 2022 Feb 1;97(2):174-184. doi: 10.1002/ajh.26397. Epub 2021 Nov 9. PMID 34724251
- [Background] Kubasch AS, Fenaux P, Platzbecker U. Development of luspatercept to treat ineffective erythropoiesis. Blood Adv. 2021 Mar 9;5(5):1565-1575. doi: 10.1182/bloodadvances.2020002177. PMID 33687432
- [Background] Attie KM, Allison MJ, McClure T, Boyd IE, Wilson DM, Pearsall AE, Sherman ML. A phase 1 study of ACE-536, a regulator of erythroid differentiation, in healthy volunteers. Am J Hematol. 2014 Jul;89(7):766-70. doi: 10.1002/ajh.23732. Epub 2014 Apr 26. PMID 24715706
- [Background] Suragani RN, Cadena SM, Cawley SM, Sako D, Mitchell D, Li R, Davies MV, Alexander MJ, Devine M, Loveday KS, Underwood KW, Grinberg AV, Quisel JD, Chopra R, Pearsall RS, Seehra J, Kumar R. Transforming growth factor-beta superfamily ligand trap ACE-536 corrects anemia by promoting late-stage erythropoiesis. Nat Med. 2014 Apr;20(4):408-14. doi: 10.1038/nm.3512. Epub 2014 Mar 23. PMID 24658078
- [Background] Markham A. Luspatercept: First Approval. Drugs. 2020 Jan;80(1):85-90. doi: 10.1007/s40265-019-01251-5. PMID 31939073
- [Background] Fenaux P, Platzbecker U, Mufti GJ, Garcia-Manero G, Buckstein R, Santini V, Diez-Campelo M, Finelli C, Cazzola M, Ilhan O, Sekeres MA, Falantes JF, Arrizabalaga B, Salvi F, Giai V, Vyas P, Bowen D, Selleslag D, DeZern AE, Jurcic JG, Germing U, Gotze KS, Quesnel B, Beyne-Rauzy O, Cluzeau T, Voso MT, Mazure D, Vellenga E, Greenberg PL, Hellstrom-Lindberg E, Zeidan AM, Ades L, Verma A, Savona MR, Laadem A, Benzohra A, Zhang J, Rampersad A, Dunshee DR, Linde PG, Sherman ML, Komrokji RS, List AF. Luspatercept in Patients with Lower-Risk Myelodysplastic Syndromes. N Engl J Med. 2020 Jan 9;382(2):140-151. doi: 10.1056/NEJMoa1908892. PMID 31914241
- [Background] Feld J, Navada SC, Silverman LR. Myelo-deception: Luspatercept & TGF-Beta ligand traps in myeloid diseases & anemia. Leuk Res. 2020 Oct;97:106430. doi: 10.1016/j.leukres.2020.106430. Epub 2020 Jul 30. PMID 32763582
- [Background] Komrokji RS, Platzbecker U, Fenaux P, Zeidan AM, Garcia-Manero G, Mufti GJ, Santini V, Diez-Campelo M, Finelli C, Jurcic JG, Greenberg PL, Sekeres MA, DeZern AE, Savona MR, Shetty JK, Ito R, Zhang G, Ha X, Backstrom JT, Verma A. Luspatercept for myelodysplastic syndromes/myeloproliferative neoplasm with ring sideroblasts and thrombocytosis. Leukemia. 2022 May;36(5):1432-1435. doi: 10.1038/s41375-022-01521-4. Epub 2022 Feb 26. No abstract available. PMID 35220402